CLINICAL TRIAL: NCT05419817
Title: Pembrolizumab With Sitravatinib in Recurrent Endometrial Cancer and Other Solid Tumors With Deficient Mismatch Repair System Post PD1 Exposure: Phase II Trial
Brief Title: Pembrolizumab With Sitravatinib in Recurrent Endometrial Cancer and Other Solid Tumors With Deficient Mismatch Repair System
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Haider Mahdi (Other)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Haider Mahdi, Assistant Professor, Department of Obstetrics, Gynecology & Reproductive Sciences, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-192
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Recurrent Endometrial Cancer; Solid Tumors
Keywords: deficient mismatch repair system (dMMR); VEGFR and KIT inhibition; anti-PD-1 therapy; checkpoint blockade
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab; sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Sitravatinib (Experimental): Standard of care pembrolizumab 200 mg IV combined with oral sitravatinib 100 mg oral QD every 21 days until disease progression, unacceptable toxicities or complete response.
  Interventions: Drug: pembrolizumab; Drug: Sitravatinib

INTERVENTIONS:
Drug: pembrolizumab — Pembrolizumab is an immunotherapy (monoclonal antibodies) that will be given at a dosage of 200 mg IV, on Day 1 of each 21 day treatment cycle
  Other Names: Keytruda®
Drug: Sitravatinib — A small molecule inhibitor of multiple tyrosine kinases that will be taken at a dosage of 100 mg orally, every day

SUMMARY:
This is a study of pembrolizumab in combination with sitravatinib in adult women with recurrent endometrial cancer or other solid tumors with deficient mismatch repair system. All patients enrolled will receive pembrolizumab as standard of care combined with Sitravatinib, which will be self-administered orally daily.

DETAILED DESCRIPTION:
This trial hypothesizes that adding anti-angiogenesis therapy to anti-PD1 therapy will reverse PD1 resistance and improve response to immunotherapy with immune checkpoint inhibitors in patients with recurrent endometrial cancer with deficient mismatch repair system. All patients enrolled will receive pembrolizumab as standard of care combined with Sitravatinib, which will be self-administered orally daily at 100 mg. Treatment will continue until disease progression or unacceptable toxicities. For patients with a complete response to therapy, maintenance therapy with both drugs will be continued for 12 months after achieving complete response. The combination of pembrolizumab with sitravatinib is an attractive treatment approach for this patient population. Sitravatinib is an orally-available, potent small molecule inhibitor of a closely related spectrum of receptor tyrosine kinases (RTKs) including MET, Axl, MERTK, VEGFR family, PDGFR family, KIT, FLT3, Trk family, RET, DDR2, and selected Eph family members. In addition to the immunostimulatory effects of Axl and MET inhibition, sitravatinib may further condition the TME in favor of antitumor activity by its immunomodulatory effects mediated through VEGFR and KIT inhibition.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment:

1. Subjects must have recurrent endometrial cancer or other solid tumors with deficient mismatch repair system. Mismatch repair deficiency is defined by 1. Immunohistochemistry with loss of expression of one of these proteins in tumor tissue as defined by standard of care: MLH1, MSH2, MSH6 and PMS2, 2. Microstaellite (MSI) unstable by PCR per standard of care, 3. MSI high by next generation sequencing using commercial platform specifically CARIS, TEMPUS or Foundation testing.
2. Must have had prior therapy with a PD1 inhibitor, pembrolizumab or other PD1/PDL1 inhibitor with confirmed radiographic progression of disease while on pembrolizumab or other PD1/PDL1 therapy.
3. Up to 5 prior lines of therapy are allowed.
4. Prior anti-angiogenesis therapy is not allowed except for bevacizumab. Prior therapy with bevacizumab is allowed.
5. Subjects must have measurable disease based on RECIST 1.1 with at least one target lesion.
6. Subjects must have an ECOG performance status of 0-1.
7. Subjects must be age >18 years. Because no dosing or adverse event data are currently available on the use of pembrolizumab in combination with sitravatinib in subjects ≤18 years of age, children are excluded from this study.
8. Subjects must have normal organ and marrow function as defined below within 14 days of enrollment unless otherwise indicated:

   * Hemoglobin ≥ 9.0 g/dl (may have been transfused)
   * Absolute neutrophil count ≥ 1,500/mcL
   * Platelet count ≥ 100,000/mcL
   * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN) range
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN orAST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
   * Estimated Creatinine clearance ≥ 40 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
   * TSH within normal institutional limits. If elevated, patient can be eligible if evaluated by an endocrine specialist, placed on replacement therapy and deemed eligible with no current or prior autoimmune disease.
9. Subjects must have the ability to understand and the willingness to sign a written informed consent document.
10. Negative serum or urine pregnancy test at screening for women of childbearing potential.
11. Willing to use highly effective contraception throughout the study and for at least 6 months after last treatment administration if childbearing potential exists
12. Availability of an archival FFPE tumor tissue block from primary diagnosis specimen, metastatic, or recurrent site. If an FFPE tissue block cannot be provided then 15 unstained slides (10 minimum) will be acceptable. Please refer to the laboratory manual for complete details.
13. Urinary protein <2+ by urine dipstick. If dipstick is >2+, then 24-hour urinary protein <2 g per 24 hours is required.
14. No evidence of uncontrolled hypertension as documented by 2 baseline blood pressure (BP) readings taken at least 1 hour apart whether same visit or different visits. The baseline systolic BP readings must be <140 mm Hg, and the baseline diastolic BP readings must be <90 mm Hg. The use of antihypertensive medications to control BP is allowed.
15. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment are eligible for this trial.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment.

1. Patients with sarcoma or carcinosarcoma
2. Mismatch repair proficient tumors
3. Prior anti-cancer therapy within 3 weeks prior to study enrollment.
4. Prior surgery or radiation within 3 weeks prior to study enrollment. Cancer directed surgery or radiation are not allowed during treatment.
5. Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable with evidence of no disease progression for 6 months.
6. Patients having received prior therapy with CTLA4 inhibitors or other immunotherapeutic agents except pembrolizumab or other anti-PD1/PDL1 therapy.
7. Patients having received prior anti-angiogenesis therapy (anti-VEGF therapy). Prior bevacizumab therapy is allowed.
8. Bowel obstruction (with or without gastrostomy tube) or inability to take oral medications
9. Patients with a prior or current bowel perforation or fistula
10. Uncontrolled hypertension defined as 140/90mmHg or greater despite medical management with multiple medications
11. Active autoimmune disease that might deteriorate when receiving an immune-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
12. Patients currently on immunosuppressive therapy except:

    * Intra-nasal, inhaled, topical or local steroid injections (e.g., intra-articular injection)
    * Steroids as premedication for hypersensitivity reaction (e.g., CT scan premedication)."
    * Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or equivalent
13. Patients who are pregnant or breast feeding.
14. Known history of immune-mediated colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis. Patients who developed any grade 2 or more immune related toxicities that require discontinuation of prior immune checkpoint inhibition will be excluded. Patients with prior immune mediated myocarditis, CNS and ocular toxicities of any grade are excluded.
15. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication or patients with ejection fraction < 40%.
16. Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
17. Prior organ transplantation including allogenic stem-cell transplantation.
18. Active infection requiring intravenous systemic therapy. Oral antibiotic therapy is allowed.
19. Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
20. Vaccination within 4 weeks of the first dose of treatment and while on trials is prohibited except for administration of inactivated vaccines. RNA-based (such as Moderna and Pfizer COVID-19 vaccines) and viral-vector (non-replicating vaccines, such as J&J COVID-19 vaccine) are considered safe and allowed.
21. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5 Grade ≥ 3)
22. Persistent toxicity related to prior therapy (NCI CTCAE v. 5 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response | At 12 weeks
  Proportion of participants with confirmed complete response or partial response by RECIST 1.1. Per RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Clinical Benefit | Up to 5 years
  Proportion of participants with complete response, partial response and stable disease by RECIST 1.1. Per RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Progression-free survival (PFS) | Up to 5 years
  Time from first response to to treatment until documented disease progression by RECIST v1.1 or death due to any cause. Progressive Disease (PD) as defined by RECIST v1.1 for target lesions: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions, (PD): Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Duration of Response (DOR) | Up to 5 years
  Time from start of complete or partial response until documented disease progression by RECIST v1.1, or death due to any cause. Progressive Disease (PD) as defined by RECIST v1.1 for target lesions: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions, (PD): Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Overall survival (OS) | Up to 5 years
  Time from first dose of study treatment until death due to any cause.
Objective response irRECIST | At 12 weeks
  Proportion of participants with confirmed Complete Response (iCR) or Partial Response (iPR) by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST). Complete Response (iCR), which describes the complete disappearance of TL and Non-TL. All lymph nodes must be non-pathological in size (< 10 mm in SAD). Partial Response (iPR), which occurs when the tumor load of the TL is reduced by ≤30% compared to the baseline, or in the case of complete remission of the TL, when one or more Non-TL can still be distinguished.
Adverse Events Related to Treatment | Up to 5 years
  Adverse Events which occur from first day of treatment, characterized by type, grade and relatedness to treatment according to NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0, considered to be possibly, probably or definitely related to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Haider Mahdi, MD, Principal Investigator — UPMC Hillman Cancer Center

IPD SHARING:
Plan to Share IPD: No